CLINICAL TRIAL: NCT02984709
Title: Check It! 2.0: Pilot Test of a Positive Psychology Intervention for Adolescents With Type 1 Diabetes
Brief Title: Check It! 2.0: Positive Psychology Intervention for Adolescents With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Sarah Jaser, Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 161732
Record Dates: First submitted 2016-11-30; First posted 2016-12-07 (Estimated); Results first posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Type1diabetes
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Positive Psychology Intervention (Experimental): The text message group will receive the intervention components via text message. They will be instructed to think about things that make them feel good when they are struggling with diabetes management (i.e. gratitude). Also they will be instructed to think about a positive value when they are in a situation that makes it hard to check their blood sugar (i.e. Self-Affirmation). Additionally, to induce positive mood they will be texted gift cards codes valued at $5.00. Further, caregivers will be asked to provide weekly positive affirmations to their adolescents, focused on non-diabetes strengths. All adolescents will be given developmentally-appropriate diabetes education material at the time of enrollment.
  Interventions: Behavioral: Positive Psychology Intervention
- Education Group (Active Comparator): The education group will be given developmentally-appropriate diabetes education material at the time of enrollment.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Positive Psychology Intervention — Health Behavior Contract - Baseline visit Education Packet - Baseline visit Positive psychology training for teen and parents - baseline visit Parent praise reminder (text message) - one time per week (over 8 week intervention period) Teen gratitude message (text message) - every Monday (over 8 week intervention period) Teen positive value message (text message) - every Wednesday (over 8 week intervention period) Teen mood booster (text message) - every Thursday and Saturday and alternative Sundays (over 8 week intervention period) Small gift ($5 gift card code sent every 2 weeks for 8 weeks)
  Other Names: Check It 2.0
  Arms: Positive Psychology Intervention
Behavioral: Education — Health Behavior Contract - Baseline visit Education Packet - Baseline visit
  Arms: Education Group

SUMMARY:
The treatment regimen for type 1 diabetes is complex and demanding, and many adolescents have problems with adherence. The proposed study will pilot test a positive psychology intervention for adolescents with type 1 diabetes aimed at improving adherence to treatment based on feedback from the first iteration of the intervention. The potential benefits include helping adolescents achieve better glycemic control, thereby reducing the health risks and complications associated with diabetes.

DETAILED DESCRIPTION:
The proposed study has the potential to improve adherence to the diabetes regimen in adolescents with type 1 diabetes without compromising their quality of life. The potential benefits include helping adolescents achieve better glycemic control, thereby reducing the health risks and complications associated with diabetes.

The investigators will use a positive psychology framework, which emphasizes positive emotions and strengths rather than problems, to promote adherence.

Positive affect, defined as feelings that reflect pleasurable engagement with the environment (e.g., happy, cheerful,proud), have been linked with favorable health outcomes and increased adherence to medical regimens. Further, positive affect has been shown to increase people's ability to use complex coping strategies. Randomized controlled trials of positive psychology interventions have been shown to successfully increase adults' adherence to medication and physical activity recommendations. However, no studies have examined the effects of positive psychology interventions on adherence behaviors in pediatric populations. Our ongoing work suggests that positive affect in adolescents with type 1 diabetes is related to greater use of adaptive coping strategies, lower levels of family conflict, and fewer depressive symptoms, and demonstrates that a positive psychology intervention has the potential to induce positive affect in adolescents. The investigators propose to pilot test a positive psychology intervention for adolescents with type 1 diabetes. This low-cost, innovative intervention is designed to induce positive affect in adolescents (age 13-17) through tailored exercises in gratitude and self-affirmation. The investigators will also promote positive parental involvement by asking caregivers to provide positive affirmation statements to adolescents. Finally, the investigators will explore the use of technology by delivering the intervention to adolescents and sending reminders to caregivers via text message using the Twilio/REDCap system.

Blood glucose monitoring is one of the best indicators of adherence to the recommended treatment regimen for type 1 diabetes, and frequency of blood glucose monitoring is strongly related to glycemic control. Further, frequency of blood glucose monitoring has been shown to decrease with age in adolescents, and parental reminders to check blood glucose are often a source of conflict between adolescents and their parents. Therefore, blood glucose monitoring represents a specific behavior that may be the best target for adherence interventions in adolescents with type 1 diabetes.

Thus, the specific aims are as follows:

Aim 1: Adapt a positive psychology intervention for adolescents (age 13-17) with type 1 diabetes designed to increase the frequency of blood glucose monitoring. Aim 2: Evaluate the feasibility, acceptability, and preliminary efficacy of a positive psychology intervention for adolescents with type 1 diabetes and their caregivers delivered by text message with the Twilio/REDCap system. The primary outcome is glycemic control, and secondary outcomes include positive affect, coping, adherence (i.e., frequency of blood glucose monitoring), family conflict, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Adolescents will be eligible if they are:

1. between the ages of 13-17;
2. have been diagnosed with type 1 diabetes for at least 1 year;
3. have no other major health problems;
4. are not currently participating in any other intervention studies;
5. have a glycosylated hemoglobin level between 7.5 - 12% on date of enrollment;
6. are patients of the Eskind Diabetes Clinic
7. must read and write in English
8. and must live the caregiver that is participating in the study with them

Exclusion Criteria:

-

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2016-10; Primary Completion 2017-02-24 (Actual); Study Completion 2017-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Jaser, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Positive Psychology Intervention: Adolescents randomized to the positive psychology group will receive the intervention components via text message. They will be instructed to think about things that make them feel good when they are struggling with diabetes management (i.e. gratitude). Also they will be instructed to think about a positive value when they are in a situation that makes it hard to check their blood sugar (i.e. Self Affirmation). Additionally, to induce positive mood they will be texted gift cards codes valued at $5.00. Further, caregivers will be asked to provide weekly positive affirmations to their adolescents, focused on non-diabetes strengths. All adolescents will be given developmentally-appropriate diabetes education material at the time of enrollment.
- Active Comparator: Education Group: Adolescents randomized to the education group will be given developmentally appropriate diabetes education material at the time of enrollment.
Period: Overall Study
Arm/Group | Experimental: Positive Psychology Intervention | Active Comparator: Education Group
Started | 24 (We enrolled 24 adolescent-parent dyads.) | 24 (We enrolled 24 adolescent-parent dyads.)
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Positive Psychology Intervention: The text message group will receive the intervention components via text message. They will be instructed to think about things that make them feel good when they are struggling with diabetes management (i.e. gratitude). Also they will be instructed to think about a positive value when they are in a situation that makes it hard to check their blood sugar (i.e. SelfAffirmation). Additionally, to induce positive mood they will be texted gift cards codes valued at $5.00. Further, caregivers will be asked to provide weekly positive affirmations to their adolescents, focused on non-diabetes strengths. All adolescents will be given developmentally-appropriate diabetes education material at the time of enrollment.
- Active Comparator: Education Group: The education group will be given developmentally appropriate diabetes education material at the time of enrollment.
- Total: Total of all reporting groups
Arm/Group | Experimental: Positive Psychology Intervention | Active Comparator: Education Group | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 24 | 24 | 48
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.0 (1.3) | 14.4 (1.2) | 14.7 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 10 | 13 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 22 | 19 | 41
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48
Glycemic Control (A1C) [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 8.60 (0.86) | 9.00 (1.07) | 8.81 (0.99)
Positive Affect [Mean (Standard Deviation); unit: score on a scale] — Positive affect measured using the Positive and Negative Affect Scale for children (PANAS-C). The positive affect scale consists of 15 items, which are summed for a total score, ranging from 15-60. Higher scores indicate higher levels of positive affect.
  score on a scale | 40.3 (7.9) | 41.2 (9.0) | 40.8 (8.4)
Frequency of Blood Glucose Monitoring [Mean (Standard Deviation); unit: number of blood glucose checks] | 3.5 (1.4) | 3.2 (1.4) | 3.2 (1.4)
Diabetes Family Conflict Scale [Mean (Standard Deviation); unit: score on a scale] — Diabetes-specific family conflict was measured with the Revised Diabetes Family Conflict Scale (DRCS), which consists of 19 items regarding how much adolescents and parents argue about diabetes management tasks. Scores range from 19-57, and higher scores indicate greater family conflict.
  score on a scale
    Parent | 24.1 (4.3) | 30 (9.1) | 27.2 (7.8)
    Teen | 30 (12) | 33 (12) | 32 (12)
Quality of Life [Mean (Standard Deviation); unit: score on a scale] — Pediatric Quality of Life Diabetes-Specific Module (PedsQL) measures quality of life. A mean scaled score is calculated, ranging from 0-100, with higher values indicating better quality of life.
  score on a scale | 70 (13) | 72 (11) | 71 (12)
Primary Control Coping [Mean (Standard Deviation); unit: ratio score] — Responses to Stress Questionnaire measures coping with diabetes-related stress. Three factors of coping are measured: primary control coping, secondary control coping,and disengagement coping. A ratio score is calculated to determine the ratio of each type of coping in relation to total coping, ranging from 0.00 to 1.00. Higher scores indicate greater relative use of primary control coping (e.g., problem solving, emotional modulation).
  ratio score | .17 (.04) | .18 (.04) | .18 (.04)
Secondary Control Coping [Mean (Standard Deviation); unit: ratio score] — Responses to Stress Questionnaire measures coping with diabetes-related stress. Three factors of coping are measured: primary control coping, secondary control coping,and disengagement coping. A ratio score is calculated to determine the ratio of each type of coping in relation to total coping, ranging from 0.00 to 1.00. Higher levels indicate greater relative use of secondary control coping (e.g., acceptance, distraction, positive thinking).
  ratio score | .26 (.05) | .27 (.05) | .27 (.05)
Disengagement Coping [Mean (Standard Deviation); unit: ratio score] — Responses to Stress Questionnaire measures coping with diabetes-related stress. Three factors of coping are measured: primary control coping, secondary control coping,and disengagement coping. A ratio score is calculated to determine the ratio of each type of coping in relation to total coping, ranging from 0.00 to 1.00. Higher levels indicate greater relative use of disengagement coping (e.g., avoidance, denial).
  ratio score | .15 (.03) | .15 (.03) | .15 (.03)
Self Care Inventory [Mean (Standard Deviation); unit: score on a scale] — The Self Care Inventory measures adherence to the recommended diabetes treatment regimen. Adolescents and parents report on the adolescents' self-care behaviors. Items are summed for a total score, ranging from 7-35. Higher scores indicate higher levels of adherence.
  score on a scale
    Parent | 24.8 (4.2) | 24.5 (4.6) | 24.7 (4.4)
    Teen | 24.8 (5.2) | 25.0 (5.1) | 24.9 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Control (A1C)
Description: A1C is the percentage of glycosylated hemoglobin and represents an average of glycemic control over the previous 2-3 months.
Time Frame: 3 months
Population: One participant in the Active Comparator group did not return for a clinic visit and therefore did not have an A1C value at follow-up.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Experimental: Positive Psychology Intervention | Active Comparator: Education Group
Number analyzed (Participants) | 24 | 23
percentage of glycosylated hemoglobin | 8.60 (1.49) | 9.35 (1.39)
Statistical Analysis 1: Comparison: Experimental: Positive Psychology Intervention; Test type: Superiority; p = 0.593, Multiple linear regression — The following a priori selected covariates were adjusted in each analysis: age, sex, race/ethnicity, income, baseline depressive symptoms, pump use, and baseline measurement for each outcome; Estimated Mean Difference = -0.170, 95% CI 2-sided [-0.81 to 0.47]

2. Secondary Outcome: Positive Affect
Description: Positive affect measured using the Positive and Negative Affect Scale for children (PANAS-C). The positive affect scale consists of 15 items, which are summed for a total score, ranging from 15-60. Higher scores indicate higher levels of positive affect.
Time Frame: 3 months
Population: One teen participant in the Experimental group did not complete follow-up survey data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Positive Psychology Intervention | Active Comparator: Education Group
Number analyzed (Participants) | 23 | 24
score on a scale | 40.6 (7.1) | 42.8 (9.2)
Statistical Analysis 1: Comparison: Experimental: Positive Psychology Intervention; Test type: Superiority; p = 0.581, Multiple linear regression — [p-value comment as in outcome 1, analysis 1]; Estimated Mean Difference = -1.137, 95% CI 2-sided [-5.27 to 2.99]

3. Secondary Outcome: Frequency of Blood Glucose Monitoring
Description: Glucometer download to determine frequency of blood glucose checks per day. Higher numbers indicates more frequent blood glucose checks.
Time Frame: 3 months
Population: Three participants in the Experimental group and five participants in the Active Comparator group did not bring their glucometers to clinic visits and therefore frequency of blood glucose monitoring could not be obtained.
Measure: Mean (Standard Deviation); unit: blood glucose checks per day
Arm/Group | Experimental: Positive Psychology Intervention | Active Comparator: Education Group
Number analyzed (Participants) | 21 | 19
blood glucose checks per day | 3.8 (1.3) | 3.2 (1.5)
Statistical Analysis 1: Comparison: Experimental: Positive Psychology Intervention; Test type: Superiority; p = 0.206, Multiple linear regression — [p-value comment as in outcome 1, analysis 1]; Estimated Mean Difference = -0.587, 95% CI 2-sided [-1.52 to 0.34]

4. Secondary Outcome: Diabetes Family Conflict Scale
Description: Diabetes-specific family conflict was measured with the Revised Diabetes Family Conflict Scale (DRCS), which consists of 19 items regarding how much adolescents and parents argue about diabetes management tasks. Scores range from 19 to 57, and higher scores indicate greater family conflict.
Time Frame: 3 months
Population: One teen participant in the Experimental group did not complete follow-up survey data. All parents completed the follow-up surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Positive Psychology Intervention | Active Comparator: Education Group
Number analyzed (Participants) | 24 | 24
score on a scale
  Diabetes Family Conflict - Teen: number analyzed (Participants) | 23 | 24
  Diabetes Family Conflict - Teen | 30 (12) | 36 (12)
  Diabetes Family Conflict - Parent | 23.8 (5.7) | 30.4 (9.6)
Statistical Analysis 1: Comparison: Experimental: Positive Psychology Intervention; Child-reported family conflict; Test type: Superiority; p = 0.511, Multiple linear regression — [p-value comment as in outcome 1, analysis 1]; Estimated Mean Difference = -2.494, 95% CI 2-sided [-10.11 to 5.13]
Statistical Analysis 2: Comparison: Experimental: Positive Psychology Intervention; Parent-reported family conflict; Test type: Superiority; p = 0.190, Multiple linear regression — [p-value comment as in outcome 1, analysis 1]; Estimated Mean Difference = -3.354, 95% CI 2-sided [-8.44 to 1.73]

5. Secondary Outcome: Diabetes-Specific Quality of Life
Description: Pediatric Quality of Life Diabetes-Specific Module (PedsQL) measures quality of life. A mean scaled score is calculated, ranging from 0-100, with higher values indicating better quality of life.
Time Frame: 3 months
Population: One teen participant in the Experimental group did not complete follow-up survey data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Positive Psychology Intervention | Active Comparator: Education Group
Number analyzed (Participants) | 23 | 24
score on a scale | 71 (14) | 71 (11)
Statistical Analysis 1: Comparison: Experimental: Positive Psychology Intervention; Test type: Superiority; p = 0.873, Multiple linear regression — [p-value comment as in outcome 1, analysis 1]; Estimated Mean Difference = 0.396, 95% CI 2-sided [-4.57 to 5.36]

6. Secondary Outcome: Primary Control Coping
Description: Responses to Stress Questionnaire measures coping with diabetes-related stress. Three factors of coping are measured: primary control coping, secondary control coping,and disengagement coping. A ratio score is calculated to determine the ratio of each type of coping in relation to total coping, ranging from 0.00 to 1.00. Higher scores indicate greater relative use of primary control coping (e.g., problem solving, emotional modulation).
Time Frame: 3 months
Population: One teen participant in the Experimental group did not complete follow-up survey data.
Measure: Mean (Standard Deviation); unit: ratio score
Arm/Group | Experimental: Positive Psychology Intervention | Active Comparator: Education Group
Number analyzed (Participants) | 23 | 24
ratio score | .18 (.03) | .20 (.04)
Statistical Analysis 1: Comparison: Experimental: Positive Psychology Intervention; Test type: Superiority; p = 0.603, Multiple linear regression — [p-value comment as in outcome 1, analysis 1]; Estimated Mean Difference = 2.996, 95% CI 2-sided [-8.57 to 14.56]

7. Secondary Outcome: Secondary Control Coping
Description: Responses to Stress Questionnaire measures coping with diabetes-related stress. Three factors of coping are measured: primary control coping, secondary control coping,and disengagement coping. A ratio score is calculated to determine the ratio of each type of coping in relation to total coping, ranging from 0.00 to 1.00. Higher levels indicate greater relative use of secondary control coping (e.g., acceptance, distraction, positive thinking).
Time Frame: 3 months
Population: One teen participant in the Experimental group did not complete follow-up survey data.
Measure: Mean (Standard Deviation); unit: ratio score
Arm/Group | Positive Psychology Intervention | Education Group
Number analyzed (Participants) | 23 | 24
ratio score | .27 (.05) | .28 (.04)

8. Secondary Outcome: Disengagement Coping
Description: Responses to Stress Questionnaire measures coping with diabetes-related stress. Three factors of coping are measured: primary control coping, secondary control coping,and disengagement coping. A ratio score is calculated to determine the ratio of each type of coping in relation to total coping, ranging from 0.00 to 1.00. Higher levels indicate greater relative use of disengagement control coping (e.g., avoidance, denial).
Time Frame: 3 months
Population: One teen participant in the Experimental group did not complete follow-up survey data.
Measure: Mean (Standard Deviation); unit: ratio score
Arm/Group | Positive Psychology Intervention | Education Group
Number analyzed (Participants) | 23 | 24
ratio score | .14 (.03) | .14 (.03)

9. Secondary Outcome: Self Care Inventory
Description: The Self Care Inventory measures adherence to the recommended diabetes treatment regimen. Adolescents and parents report on the adolescents' self-care behaviors. Items are summed for a total score, ranging from 7-35. Higher scores indicate higher levels of adherence.
Time Frame: 3 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Positive Psychology Intervention | Education Group
Number analyzed (Participants) | 23 | 24
score on a scale
  Self Care Inventory - Parent | 26.6 (3.9) | 25.9 (5.2)
  Self Care Inventory - Teen | 25.2 (5.1) | 26.0 (5.3)

ADVERSE EVENTS:
Time Frame: 1 year
Description: We do not anticipate that any adverse events will arise from study participation, as this is a behavioral intervention. Normal blood glucose management, including treatment of hypoglycemia, is a standard practice in diabetes management and would not be considered an adverse event.
Arm/Group | Experimental: Positive Psychology Intervention | Active Comparator: Education Group
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT02984709/SAP_000.pdf
  • Study Protocol (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT02984709/Prot_001.pdf